CLINICAL TRIAL: NCT02500277
Title: A Study to Evaluate the Yield of Pleural Biopsy With a Flexible Cryoprobe Versus Flexible Forceps During Semirigid Thoracoscopy: a Comparative Study
Brief Title: Yield of Cryoprobe vs Flexible Forceps Pleural Biopsy
Acronym: COFFEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NK/1815/Res/2439
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pleural Effusion; Pleurisy; Tuberculosis; Metastatic Malignancy
Keywords: thoracoscopy; pleuroscopy; semirigid thoracoscopy; flexible cryoprobe; cryobiopsy; pleural biopsy
MeSH Terms: conditions — Pleural Effusion; Pleurisy; Tuberculosis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryobiopsy (Active Comparator): Pleural biopsy with a flexible cryoprobe
  Interventions: Device: Cryoprobe pleural biopsy first
- Forceps biopsy (Active Comparator): Pleural biopsy with a flexible forceps
  Interventions: Device: Flexible forceps biopsy first

INTERVENTIONS:
Device: Cryoprobe pleural biopsy first — Four pleural biopsy specimens will be obtained using the flexible cryoprobe (ERBOCRYOCA, ERBE, Tubingen, Germany; outer diameter 1.9 mm, length 900 mm) followed by 6-10 pleural biopsy specimens obtained using the flexible thoracoscopic forceps (FB-55CR, Olympus Medical Systems, 2 mm diameter).
  Arms: Cryobiopsy
Device: Flexible forceps biopsy first — Six to ten pleural biopsy specimens will be obtained using the flexible thoracoscopic forceps (FB-55CR, Olympus Medical Systems, 2 mm diameter) followed by four pleural biopsy specimens obtained using the flexible cryoprobe (ERBOCRYOCA, ERBE, Tubingen, Germany; outer diameter 1.9 mm, length 900 mm)
  Arms: Forceps biopsy

SUMMARY:
This is a prospective study to assess the yield of pleural biopsy obtained with the routine flexible thoracoscopic biopsy forceps versus that obtained with a flexible cryoprobe during semirigid thoracoscopy

DETAILED DESCRIPTION:
Consecutive patients with exudative pleural effusions who are planned to undergo semirigid thoracoscopy will be enrolled in the study if they satisfy the inclusion criteria. They will be randomized in 1:1 ratio using a computer-generated randomization sequence to the following groups:

Group A: Four pleural biopsy specimens obtained using the flexible cryoprobe followed by eight pleural biopsy specimens obtained using the flexible thoracoscopic forceps OR Group B: The above two procedures will be performed in the reverse order The biopsies will be performed from different areas of the involved pleura with the two techniques. Thoracoscopy will be performed in the bronchoscopy suite on spontaneously breathing subjects (fasting for 8 h) under conscious sedation (using midazolam, pentazocine, and tramadol) observing complete aseptic precautions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years
* Semirigid thoracoscopy being performed for diagnosis of the pleural effusion

Exclusion Criteria:

* Age ≥80 years
* SpO2 <88% on room air
* Hemodynamic instability
* Myocardial infarction or unstable angina in the last 6 wk
* Lack of pleural space due to adhesions
* Uncorrected coagulopathy
* Failure to provide informed consent

Ages: 12 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Yield of pleural biopsy obtained with the routine flexible thoracoscopic biopsy forceps versus that obtained with a flexible cryoprobe during semirigid thoracoscopy | One week
  The proportion of patients where a definitive histopathological diagnosis was obtained will be compared between the cryoprobe and flexible forceps biopsy

SECONDARY OUTCOMES:
Biopsy size | One day
  Size of biopsy specimens obtained with the two techniques
Duration of procedure | One day
  Time taken for the procedure with the two techniques
Ease of biopsy VAS | One day
  Ease of taking biopsy with the two techniques assessed using a visual analog scale
Artifacts | One day
  Number of patient speciemens with histopathologic artifacts with either technique including crush artefacts with the flexible forceps and freeze artifacts with the cryoprobe
Tissue depth | One day
  Depth of the tissue obtained on histopathology
Bleeding | One day
  Number of participants with bleeding seen while taking biopsy categorised into "no bleeding", "minimal self limited ooze", "bleeding requiring prolonged suctioning" , "major hemorrhage requiring blood transfusion, causing hemodynamic instability or ICU admission"

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India